CLINICAL TRIAL: NCT03304704
Title: Community Dynamics of Malaria Transmission and Mosquito Feeding in Bancoumana and Doneguebougou, Mali
Brief Title: Community Dynamics of Malaria Transmission and Mosquito Feeding in Bancoumana, Mali
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999917180; 17-I-N180
Record Dates: First submitted 2017-10-06; First posted 2017-10-09 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Malaria
Keywords: Assays; Direct Skin Feeds; Infection; Parasite; Gametocyte; Natural History
MeSH Terms: conditions — Malaria; Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- DSF Cohort: Accrual/Screening up to 1800 will include volunteers between the ages of 5 and 17 years and will be enrolled for genotyping and monthly blood sampling
- Genotype Cohort: Accrual/Screening up to 1500 will complete a single visit with blood draw for genotyping for future fidelity assessments with blood-fed, spray wild-caught mosquitoes.
- Parasite Surveillance Cohort: Accrual/Screening up to 1500 will be enrolled for genotyping and a minimum of six monthly blood sampling and mosquito wild catches wild-caught mosquitoes within their compound

SUMMARY:
Background:

Half of the world's population is at risk of malaria. Malaria is a disease that affects many people in Mali and other parts of Africa. It is caused by germs spread by mosquito bites. Malaria may be mild. But it can also be serious or can lead to death if it is not diagnosed and treated promptly. Researchers want to learn more about the disease so they can develop new approaches to malaria control.

Objective:

To collect data on how mosquitoes spread malaria and how many people get malaria in the community by comparing different areas, seasons, and years.

Eligibility:

Residents of a certain area of Mali who are of any age

Design:

Participants will be screened with a physical exam and medical history.

All participants will have at least 1 visit. They will answer questions about their health and malaria. They may have a physical exam. They will have blood collected.

Some participants will have 1 visit every month for 3 years. They will repeat the procedures above.

These participants will have mosquitoes collected in their home monthly. They may be able to catch some of the mosquitoes alive or may need to use a spray to kill the mosquitoes. Participants in this part of the study can be up to 65 years old.

Some participants will also have about 60 mosquitoes directly feed on their arm or leg for 15-20 minutes each month. These participants must be 5-65 years old.

...

DETAILED DESCRIPTION:
A vaccine that interrupts malaria transmission is critical to eradicate the disease, but improved assays are needed to measure the efficacy of vaccines. Transmission-blocking vaccines (TBVs) work by inducing antibodies in vaccinees that inhibit parasite development in the mosquito interrupting transmission. Efficacy of vaccines may be estimated by in vitro membrane feeding assays using immune sera and laboratory mosquitoes, but qualified assays that measure transmission in the field are needed to assess transmission-blocking interventions in natura. Clinical trials of TBV have started in Bancoumana and Doneguebougou, and we expect to expand TBV studies here and in adjacent areas in the future. This protocol will use a longitudinal cohort to gather information on mosquito feeding and infection patterns in Bancoumana, Doneguebougou and surrounding villages in Mali. Individuals actively participating in LMIV vaccine trials will be approached first for participation, including permission to contact their household and neighbors of their compound for participation. Households will be identified using census data and individuals will be consented for participation. Malaria smears will be obtained at monthly visits, in conjunction with mosquito collections in/around village residences and with direct skin feeds (DSFs) using insectary-raised mosquitoes. Parasite transmission to mosquitoes will be assessed longitudinally for differences by season and year, and compared between wild-caught and laboratory-raised mosquitoes. Data will also be obtained on gametocyte and parasite carriage rates by season and year. Genotyping of individual subjects will be performed to pair with the bloodmeals of wild-caught mosquitoes.

A total of 3,200 volunteers from Bancoumana, Doneguebougou and surrounding areas will be enrolled into three distinct cohorts. The Genotype Only Cohort (n=1000), which will include the vaccine trial participants, will complete a single visit to obtain a blood sample for genotyping with no additional follow up. The DSF Cohort (n=1200) will enroll subjects aged 5 to 65 years for monthly blood sampling, DSF, and mosquito collection at their household. The Parasite Surveillance Cohort (n=1000) will enroll subjects under the age of 5 years (as young as 6 months) and subjects of any age who are unwilling to participate in DSF; they will have monthly blood sampling and mosquito collection at their household. Enrollment into the Genotype and Parasite Surveillance Cohorts will be linked to full enrollment of the DSF Cohort. Participants in the Parasite Surveillance and DSF cohorts, will be followed for up to 3 years, to collect data that will guide the design of future community-based trials of TBV.

ELIGIBILITY:
* INCLUSION CRITERIA:
* GENOTYPE ONLY COHORT

  * Any age
  * Known resident of Bancoumana or the surrounding villages
  * Acceptance and signature of the written informed consent and the assent for children aged 12-17 years
  * Willingness to allow stored laboratory specimens to be used for future research
* PARASITE SURVEILLANCE COHORT

  * 6 months to 65 years of age
  * Known resident of Bancoumana or the surrounding villages
  * Willingness to allow stored laboratory specimens to be used for future research
  * Acceptance and signature of the written informed consent and the assent for children aged 12-17 years
* DSF COHORT

  * Aged between 5 and 65 years, inclusive
  * Good general health as determined by review of medical history and/or clinical testing at the time of screening
  * Known resident of Bancoumana or the surrounding villages
  * Willingness to allow stored laboratory specimens to be used for future research
  * Willingness to undergo DSF
  * Acceptance and signature of the written informed consent and the assent for children aged 12-17 years

EXCLUSION CRITERIA:

* GENOTYPE ONLY COHORT

  * Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol
  * Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol
* PARASITE SURVEILLANCE CHORT

  * Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol
  * Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol
  * Currently enrolled participant in protocol 17-I-N006 or another active LMIV/MRTC vaccine clinical trial
* DSF COHORT

  * Behavioral, cognitive, or psychiatric disease that in the opinion of the investigator affects the ability of the subject to understand and cooperate with the study protocol
  * Other condition that, in the opinion of the investigator, would jeopardize the safety or rights of a volunteer participating in the trial or would render the subject unable to comply with the protocol
  * Currently enrolled participant in protocol 17-I-N006 or another LMIV/MRTC vaccine clinical trial
  * History of severe reaction to mosquito bites

Ages: 6 Months to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Known resident of Bancoumana, Doneguebougou or the surrounding villages; and Willingness to allow stored laboratory specimens to be used for future research@@@@@@
Sampling Method: Non-Probability Sample
Enrollment: 1928 (Actual)
Dates: Start 2018-01-28 (Actual); Primary Completion 2020-07-12 (Actual); Study Completion 2020-07-12 (Actual)

PRIMARY OUTCOMES:
Measurement of estimated rates of Infection rate in mosquitoes by DSF measured as the rate (per blood-fed mosquito) of malaria transmission (human to mosquito) | Up to 3 years
  Infection rate in mosquitoes by DSF measured as the rate (per blood-fed mosquito) of malaria transmission (human to mosquito; and Infection rate in live wild-caught mosquitoes measured as the rate (per blood-fed mosquito) of malaria transmission (human to mosquito)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer C Hume, Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (3):
- Mali (3):
  - Bancoumana Malaria Vaccine Center, Bamako
  - Univ of Sciences, Techniques and Technology, Bamako
  - Doneguebougou Facility, Donéguébougou

REFERENCES:
- [Background] Toure YT, Doumbo O, Toure A, Bagayoko M, Diallo M, Dolo A, Vernick KD, Keister DB, Muratova O, Kaslow DC. Gametocyte infectivity by direct mosquito feeds in an area of seasonal malaria transmission: implications for Bancoumana, Mali as a transmission-blocking vaccine site. Am J Trop Med Hyg. 1998 Sep;59(3):481-6. doi: 10.4269/ajtmh.1998.59.481. PMID 9749648
- [Background] Diallo M, Toure AM, Traore SF, Niare O, Kassambara L, Konare A, Coulibaly M, Bagayogo M, Beier JC, Sakai RK, Toure YT, Doumbo OK. Evaluation and optimization of membrane feeding compared to direct feeding as an assay for infectivity. Malar J. 2008 Dec 2;7:248. doi: 10.1186/1475-2875-7-248. PMID 19055715
- [Background] Drakeley C, Sutherland C, Bousema JT, Sauerwein RW, Targett GA. The epidemiology of Plasmodium falciparum gametocytes: weapons of mass dispersion. Trends Parasitol. 2006 Sep;22(9):424-30. doi: 10.1016/j.pt.2006.07.001. Epub 2006 Jul 17. PMID 16846756